CLINICAL TRIAL: NCT01523457
Title: Phase II Study of Modified FOLFIRINOX in Advanced Pancreatic Cancer
Brief Title: Study of Modified FOLFIRINOX in Advanced Pancreatic Cancer
Acronym: FOLFIRINOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1108008901
Record Dates: First submitted 2012-01-23; First posted 2012-02-01 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-05

CONDITIONS: Metastatic Pancreatic Cancer; Pancreatic Cancer
Keywords: metastatic pancreatic cancer; locally advanced pancreatic cancer; FOLFIRINOX; phase II; progression free survival
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MPC modified FOLFIRINOX (Experimental): Patients with metastatic pancreatic cancer (MPC) were treated with modified FOLFIRINOX every 2 weeks as follows: oxaliplatin 85 mg m 2 infused over 120 min, immediately followed by folinic acid 400 mg m 2 infused over 120 min with the addition, after 30 min, of irinotecan 135 mg m 2 infused over 90 min, followed by 5FU 300 mg m 2 IV bolus, followed by 2400 mg m 2 continuous infusion for 46 h (25% reduction in bolus 5FU and irinotecan doses). All patients received pegylated filgrastim with each cycle on day 3 or 4 in the absence of severe leukocytosis. All patients routinely received palonosetron, aprepitant and dexamethasone for emesis prophylaxis.
  Interventions: Drug: Folfirinox
- LAPC modified FOLFIRINOX (Experimental): Patients with locally advanced pancreatic cancer (LAPC) were treated with modified FOLFIRINOX every 2 weeks as follows: oxaliplatin 85 mg m 2 infused over 120 min, immediately followed by folinic acid 400 mg m 2 infused over 120 min with the addition, after 30 min, of irinotecan 135 mg m 2 infused over 90 min, followed by 5FU 300 mg m 2 IV bolus, followed by 2400 mg m 2 continuous infusion for 46 h (25% reduction in bolus 5FU and irinotecan doses). All patients received pegylated filgrastim with each cycle on day 3 or 4 in the absence of severe leukocytosis. All patients routinely received palonosetron, aprepitant and dexamethasone for emesis prophylaxis.
  Interventions: Drug: Folfirinox

INTERVENTIONS:
Drug: Folfirinox — * Oxaliplatin 85 mg/m2 IV infused over two hours, followed by
  * Leucovorin 400 mg/m2 IV over two hours
  * Irinotecan 135 mg/m2 IV over 90 minutes (concurrent with leucovorin during the last 90 min of the leucovorin infusion)
  * 5-FU 300mg/m2 IV bolus, then 2400 mg/m2 continuous IV infusion over 46 hours
  FOLFIRINOX is a chemotherapy regimen. It is made up of the following four drugs:
  FOL - folinic acid (leucovorin), a vitamin B derivative that modulates/potentiates/reduces the side effects of fluorouracil; F - fluorouracil (5-FU), a pyrimidine analog and antimetabolite which incorporates into the DNA molecule and stops DNA synthesis; IRIN - irinotecan (Camptosar), a topoisomerase inhibitor, which prevents DNA from uncoiling and duplicating; and OX - oxaliplatin (Eloxatin), a platinum-based antineoplastic agent, which inhibits DNA repair and/or DNA synthesis.

SUMMARY:
The primary objective of this study was to determine the progression free survival in patients with metastatic pancreatic cancer and in patients with locally advanced unresectable non-metastatic pancreatic cancer treated with a dose-attenuated modification of folinic acid, fluorouracil, irinotecan, and oxaliplatin (FOLFIRINOX). Secondary endpoints included: determine objective response rate according to RECIST; determine overall survival; evaluate toxicity; determine rate of resection in locally advanced unresectable stratum; correlate time to progression, objective response, and overall survival with early changes in glucose metabolism using [18F]-fluorodeoxyglucose (FDG)-positron emission tomography (PET) scanning.

DETAILED DESCRIPTION:
A phase II open label single arm multi-institutional study at Yale's Smilow Cancer Hospital (New Haven, CT, USA), the Smilow Cancer Hospital Care Centers (regional community-based clinics), the VA Connecticut Healthcare System West Haven Campus (West Haven, CT, USA) and Bridgeport Hospital (Bridgeport, CT, USA). The primary objective of this study was to determine the PFS in patients with MPC and LAPC treated with a dose attenuated modification of FOLFIRINOX.

NOTE: Upon results reporting (2016), the registration record was reorganized to display MPC and LAPC groups in individual arms. The most meaningful comparison is between MPC/LAPC and historical controls. That is how results are reported in the published paper, see citations.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic or cytologic documentation of pancreatic adenocarcinoma
* Metastatic or locally advanced unresectable disease, including borderline unresectable disease
* Patients with biliary or gastroduodenal obstruction must have drainage or surgical bypass prior to starting chemoradiation
* Measurable or non-measurable assessable disease
* No prior treatment (chemotherapy, biological therapy, or radiotherapy) for metastatic or non-metastatic locally advanced unresectable pancreatic cancer
* 6 months since completion of any prior neoadjuvant or adjuvant therapy (chemotherapy or radiotherapy) for resected pancreatic cancer
* No prior treatment with oxaliplatin or irinotecan
* No prior treatment with fluoruouracil or capecitabine unless administered as a radiosensitizing drug during adjuvant/neoadjuvant chemoradiotherapy after/before resection of pancreatic cancer
* Patients who received chemotherapy > 2 years ago for malignancies other than pancreatic cancer are eligible, provided that chemotherapy was completed > 2 years ago and there is no evidence of the second malignancy at the time of study entry
* > 4 weeks since major surgery
* No other concurrent anticancer therapy
* ECOG Performance Status: 0-1
* Age > 18
* No other malignancy within past two years except basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer
* Paraffin block or slides must be available
* Adequate organ function
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No > grade 1 sensory peripheral neuropathy
* No uncontrolled seizure disorder, active neurological disease, or known CNS disease
* No significant cardiac disease, including the following: unstable angina, New York Heart Association class II-IV congestive heart failure, myocardial infarction within six months prior to study enrollment
* No history of chronic diarrhea
* Not pregnant and not nursing
* No other medical condition or reason that, in the opinion of the investigator, would preclude study participation
* Laboratory parameters as follows: absolute neutrophil count ≥ 1,500/uL, platelet count ≥ 100,000/uL, hemoglobin ≥ 9 g,/dL, creatinine < 1.5 X ULN or estimated GFR > 30 ml/min, bilirubin < 1.5 X ULN, AST and ALT < 3 X ULN, negative pregnancy test in women of childbearing age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Lacy, MD, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Center, New Haven, Connecticut, United States

REFERENCES:
- [Result] Stein SM, James ES, Deng Y, Cong X, Kortmansky JS, Li J, Staugaard C, Indukala D, Boustani AM, Patel V, Cha CH, Salem RR, Chang B, Hochster HS, Lacy J. Final analysis of a phase II study of modified FOLFIRINOX in locally advanced and metastatic pancreatic cancer. Br J Cancer. 2016 Mar 29;114(7):737-43. doi: 10.1038/bjc.2016.45. PMID 27022826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with pathologically confirmed, measurable or non-measurable assessable MPC or LAPC (including unresectable and borderline resectable) were recruited from November 2011 through January 2014.
Period: Overall Study
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Started | 44 | 31
Completed | 37 | 29
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Population: 75 patients, including 44 with MPC and 31 with LAPC, were enrolled. The demographics and disease characteristics of the 37 evaluable patients in the MPC cohort in this study are presented here. Seven of 44 patients with MPC were excluded from efficacy analysis due to voluntary withdrawal.
Groups:
- Total: Total of all reporting groups
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX | Total
Number analyzed (Participants) | 37 | 31 | 68
Age, Customized [Median (Full Range); unit: years]
  Age | 62 [50 to 77] | 63 [46 to 79] | 62 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 21 | 20 | 41
ECOG Performance Status [Number; unit: participants]
  0: Fully active | 17 | 15 | 32
  1: Restricted in physically strenuous activity | 20 | 16 | 36
Pancreatic tumour location [Number; unit: participants] — Location of the pancreatic tumour in either the head or body of the pancreas. Six subjects had their pancreatic tumour resected (so it is no longer located in the pancreas), but still qualified for the metastatic arm.
  participants
    Head | 17 | 27 | 44
    Body | 14 | 4 | 18
    Tumour Resection | 6 | 0 | 6
Level of CA19.9 [Number; unit: participants] — CA 19-9 (carbohydrate antigen 19-9 is a tumor marker that is used primarily in the management of pancreatic cancer. Changes in CA 19-9 levels help determine if the tumor is growing, remaining stable or getting smaller.
  participants
    Normal | 4 | 3 | 7
    Elevated, <59 Upper Limits of Normal | 18 | 24 | 42
    Elevated, >=59 Upper Limits of Normal | 15 | 4 | 19
Biliary stent [Number; unit: participants]
  Yes | 9 | 17 | 26
  No | 28 | 14 | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary objective of this study is to determine the progression free survival in patients with metastatic pancreatic cancer and in patients with locally advanced unresectable non-metastatic pancreatic cancer treated with a dose-attenuated modification of FOLFIRINOX. Tumour response was determined according to RECIST 1.1 by independent radiology review.
Time Frame: 24 weeks
Population: Two of 31 patients with LAPC were excluded from efficacy analysis because they did not complete four cycles to reach the first efficacy assessment (one due to cholecystitis with abscess and one due to cerebrovascular accident).
Measure: Number; unit: percentage of participants
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Number analyzed (Participants) | 37 | 29
percentage of participants | 54 | 97

2. Secondary Outcome: Objective Response Rate
Description: Response will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1 by independent radiology review) at 8 week intervals in patients with metastatic disease and in patients with locally advanced disease.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Number analyzed (Participants) | 37 | 29
percentage of participants | 35.1 | 17.2

3. Secondary Outcome: Overall Survival
Description: Overall survival will be determined in patients with metastatic disease and in patients with locally advanced disease.
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Number analyzed (Participants) | 37 | 29
percentage of participants | 81 | 100

4. Secondary Outcome: Toxicity
Description: Toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) 4.0. Rates of grade 3 and 4 toxicities will be compared to historical controls. MPC and LAPC are combined because they were given the exact same medication. The study aimed to compare this dosage with historical dosage, so this comparison is the most appropriate.
Time Frame: 24 weeks
Population: One of the total 75 patients did not receive treatment and was excluded from toxicity analysis. Treatment-related grade 3 and 4 adverse events observed in our study and in the historical control group treated with standard FOLFIRINOX.
Measure: Number; unit: participants
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Number analyzed (Participants) | 43 | 31
participants
  Neutropenia | 4 | 5
  Thrombocytopenia | 5 | 2
  Anaemia | 2 | 2
  Febrile neutropenia | 1 | 2
  Diarrhea | 8 | 4
  Fatigue | 5 | 4
  Alanine aminotransferase (ALT) increased | 3 | 0
  Thromboembolic event | 3 | 0
  Peripheral sensory neuropathy | 2 | 0
  Vomiting | 1 | 1

5. Secondary Outcome: Rate of Resection in Patients With Locally Advanced Disease
Description: The rate of surgical resection in the cohort of patients with locally advanced disease will be determined.
Time Frame: 24 weeks
Population: Only LAPC patients were considered in the analysis. 13 patients in the LAPC group had surgical resection. The definition of locally unresectable and borderline were clarified in the protocol.
Measure: Number; unit: participants
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Number analyzed (Participants) | 0 | 31
participants
  Total |  | 13
  Unresectable |  | 6
  Borderline |  | 7

6. Secondary Outcome: Correlate Time to Progression, Objective Response, and Overall Survival With Early Changes in Glucose Metabolism Using FDG-positron Emission Tomography (PET) Scanning
Description: The time to progression, objective response rate, and overall survival will be correlated with early changes in glucose metabolism using FDG-positron emission tomography (PET) scanning in patients with metastatic disease and locally advanced disease.
Time Frame: 24 weeks
Population: This outcome was included in the 2012 protocol registration and actually describes a series of analyses that were not fully conducted, and will not be. The outcome measures described in the outcome description are presented as separated outcome measures elsewhere in this results record.
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported over the total duration of the study by treatment arm.
Description: Reported below are grade 3 and 4 adverse events reported at greater than 5% per treatment arm collected. Serious Adverse Events and All Cause Mortality are reported for the overall population, while the Adverse Events are reported only for those where toxicity was assessed (1 less participant overall, see Outcome Measures).
Arm/Group | MPC Modified FOLFIRINOX | LAPC Modified FOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/31
Other Adverse Events (participants affected / at risk) | 20/43 | 11/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MPC Modified FOLFIRINOX (N=43) | LAPC Modified FOLFIRINOX (N=31)
Neutropenia (Blood and lymphatic system disorders) | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile Neurotropenia (Blood and lymphatic system disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 8 | 4
Fatigue (General disorders) | 5 | 4
Alanine aminotransferase (General disorders) | 3 | 0
Thromboembolic Event (Blood and lymphatic system disorders) | 3 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes